CLINICAL TRIAL: NCT02042287
Title: Controlled, Multicenter, Randomized Parallel Group Pilot Study With 2 Treatment Arms in Non-pregnant Women With Acute Symptomatic Bacterial Vaginosis (BV)
Brief Title: Treatment Comparison of Antibiotics Versus Vaginal Lactic Acid in Non-pregnant Women With Acute Symptomatic Bacterial Vaginosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Tentan AG (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 026/13
Record Dates: First submitted 2014-01-20; First posted 2014-01-22 (Estimated); Last update posted 2022-04-08 (Actual); Status verified 2022-03

CONDITIONS: Bacterial Vaginosis
Keywords: Bacterial Infections and Mycoses; Pharmaceutical Preparations; Health Occupations
MeSH Terms: conditions — Vaginosis, Bacterial; Bacterial Infections and Mycoses | interventions — Metronidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1: Gynofit® (Experimental): Vaginal lactic acid gel
  Interventions: Device: Vaginal lactic acid and glycogen gel
- 2: metronidazole (Active Comparator): Oral antibiotic
  Interventions: Drug: Metronidazole

INTERVENTIONS:
Device: Vaginal lactic acid and glycogen gel — Medical device (registration number: 10-355-717, first licensed 12.08.2010)
  Arms: 1: Gynofit®
Drug: Metronidazole — Oral antibiotic
  Arms: 2: metronidazole

SUMMARY:
Bacterial vaginosis (BV) is the most common cause of vaginitis in women of childbearing age. Women with symptomatic BV may present with malodorous discharge that is off-white, thin, and homogenous and has a fishy smell especially after intercourse. It is of importance to treat women with BV, as this condition is associated with serious risks, such as an increased risk of preterm birth in pregnant women, and particular vulnerability to the acquisition of sexually transmitted disease (STD). The pathophysiology of BV consists of changes in the microbiologic composition of the vaginal flora. The treatment of choice for BV is oral metronidazole for 7 days. Although the available antibiotic therapies produce good results in the short term, symptomatic BV persists or recurs at 3 months in up to 50% to 70% of patients, with long-term recurrence approaching 85%. An alternative treatment option may be a vaginal acid gel which aims to optimize the vaginal milieu. The aim of this pilot study is to assess the efficacy of Gynofit® vaginal gel (lactic acid and glycogen) compared to oral metronidazole in the treatment of BV.

DETAILED DESCRIPTION:
Background

Bacterial vaginosis (BV) is the most common cause of vaginitis in women of childbearing age, with an estimated prevalence of 29% in the general population of women aged 14 to 49 years.

Women with symptomatic BV may present with malodorous discharge that is off-white, thin, and homogenous and has a fishy smell especially after intercourse. However, only the minority of women with BV is symptomatic.

Regardless of the symptoms, it may be of importance to treat women with BV, as this condition is associated with serious risks, such as an increased risk of preterm birth in pregnant women, particular vulnerability to the acquisition of sexually transmitted disease (STD), including gonorrhea, chlamydia trachomatis, genital herpes and HIV and a possibly higher risk of pelvic inflammatory disease (PID). Moreover, endometrial bacterial colonization, plasma-cell endometritis, postpartum fever, post-hysterectomy vaginal cluff cellulitis and post-abortal infection seem to be associated with BV.

The pathophysiology of BV consists of changes in the microbiologic composition of the vaginal flora. In the healthy vaginal flora, lactobacilli are the predominant bacteria, producing lactic acid and H2O2, maintaining a pH<4.5 and inhibiting the growth of other organisms. In BV, the concentration of H2O2-producing lactobacilli is reduced and other species become more prevalent, notably Gardnerella vaginalis, Prevotella species, Porphyromonas species, Bacteroides species, Peptostreptococcus species, Mycoplasma hominis, Ureaplasma urealyticum, and Mobiluncus species. These vaginal anaerobes produce carboxylase enzymes, breaking down peptides to amines, which get volatile and malodorous with the increased pH. More over the amines increase vaginal transudation and squamous epithelial cell exfoliation, leading to the typical discharge in BV. With the increased pH, Gardnerella vaginalis can adhere to squamous epithelial cells and create a biofilm. The mechanism by which this floral imbalance occurs is not clear, but sexual activity seems to be a major risk factor, as BV does not occur in sexual inactive women. Additionally, multiple or new sexual partners, frequency of vaginal intercourse, vaginal douching, and cigarette smoking have also been identified as risk factors, whereas the use of condoms had a protective effect.

BV can be diagnosed by the use of clinical criteria or Gram stain. For standard clinical use, practical diagnostic criteria were proposed by Amsel et al.. Amsel criteria include: (a) an adherent grayish-white discharge; (b) a positive whiff test (a fishy odor of the vaginal discharge before or after addition of 10% potassium hydroxide); (c) an elevated vaginal pH (pH > 4.5); and (d) the presence of clue cells on microscopy. The diagnosis of BV is made, if 3 of these 4 symptoms are present.

A Gram stain (Nugent Score) is considered the gold standard laboratory method for diagnosing BV and determines the relative concentration of Gram-positive lactobacilli, Gram-negative and Gram-variable rods and cocci and curved Gram-negative rods characteristic of BV.

BV resolves spontaneously in up to one-third of non-pregnant and one-half of pregnant women. The Centers for Disease Control and Prevention (CDC) recommend a treatment for all non-pregnant women with symptomatic BV to relieve vaginal symptoms and signs of infection. Treatment is also indicated to prevent postoperative infection in those with asymptomatic infection prior to abortion or hysterectomy. Some experts recommend treating all women with BV, for reducing the risk of acquiring STDs.

The treatment of choice for BV is oral metronidazole 500 mg orally twice a day for 7 days. Other recommended regimens are metronidazole gel 0.75%, one full applicator (5 g) intravaginally, once a day for 5 days; or clindamycin cream 2%, one full applicator (5 g) intravaginally at bedtime for 7 days. Alternative regimens are tinidazole 2 g orally once daily for 2 days; or tinidazole 1 g orally once daily for 5 days; or clindamycin 300 mg orally twice daily for 7 days; or clindamycin ovules 100 mg intravaginally once a bedtime for 3 days. Oral metronidazole is considered the treatment of choice with a cure rate of 80 - 90%.

Although the available antibiotic therapies produce good results in the short term, symptomatic BV persists or recurs at 1 month in approximately 11% to 29% of patients. At 3 months, recurrence of BV has been reported in 50% to 70% of patients, with long-term recurrence approaching 85%.

Although the causes of recurrence are not known, it has been found that the vaginal biofilm with Gardnerella vaginalis and Atopobium vaginae persisted after treatment, probably explaining the high recurrence rates.

In in vitro studies lactobacilli were able to disrupt the biofilm and reduce the risk of BV. Thus, it is being investigated, if recolonizing the vagina with healthy stains of H2O2-producing lactobacilli could prevent relapse after treatment. Systemic reviews of trials investigating probiotics for treatment of BV have not found sufficient evidence for or against efficacy.

Acidification is another treatment option, as lowering the vaginal pH encourages the growth of lactobacilli. In one study, acid gel was as effective as metronidazole in the treatment of BV. Similarly, in an observational study, the use of acetic acid vaginal gel after the treatment of BV significantly reduced the rate of recurrence. However, data on the treatment and prevention efficacy by acidification is scarce and controversial.

Objective

The principal exploratory goal of the present pilot study is to assess the efficacy of Gynofit® vaginal gel (lactic acid and glycogen) compared to oral metronidazole in the treatment of BV.

Methods

In this pilot study clinical efficacy of treatment will be assessed using the Amsel criteria, which are diagnostic criteria used in standard clinical practice. The Nugent score, a laboratory method for diagnosing BV, will be measured as well to confirm clinical findings. Finally, subjective BV symptoms are assessed by means of a questionnaire to determine the subjective effectiveness of treatment.

The following collaborator is providing support for this study: Dr. rer. nat. Ulrich Stefenelli, Würzburg, Germany.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old
* Acute symptomatic BV
* Signed informed consent

Exclusion Criteria

* Insufficient knowledge of German
* Illiteracy
* Pregnancy
* Acute illness
* Known allergies against ingredients of the investigational products

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-06; Primary Completion 2020-03-19 (Actual); Study Completion 2020-03-19 (Actual)

PRIMARY OUTCOMES:
Proportion (percentage) of patients with treatment success based on the Amsel criteria at week 3. | Visit 1 (day 0) and Visit 2 (day 21)
  This is a binary parameter indicating remission from BV.

SECONDARY OUTCOMES:
Proportion (percentage) of patients with treatment success based on the Nugent score at week 3. | Visit 1 (day 0) and Visit 2 (day 21)
  This is a binary parameter indicating remission from BV.
Mean symptom score-changes (as pre-post-difference) regarding severity of BV at week 3 | Visit 1 (day 0) and Visit 2 (day 21)
  Unpleasant vaginal discharge, unpleasant smell, vaginal pain, itching, burning, dryness
Percentage of patients with a complete relief from symptoms | Visit 1 (day 0), Visit 2 (day 21), Visit 3 (day 84) and Visit 4 (day 252

CONTACTS AND LOCATIONS:
Overall Officials: Petra Stute, MD, Study Chair — Department of Obstetrics and Gynecology Inselspital Bern
Locations (1):
- Dep. of Obstetrics and Gynecology, Bern University Hospital, Bern, Bern, Switzerland

REFERENCES:
- [Background] Schwebke JR. Gynecologic consequences of bacterial vaginosis. Obstet Gynecol Clin North Am. 2003 Dec;30(4):685-94. doi: 10.1016/s0889-8545(03)00086-x. PMID 14719845
- [Background] Hill GB. The microbiology of bacterial vaginosis. Am J Obstet Gynecol. 1993 Aug;169(2 Pt 2):450-4. doi: 10.1016/0002-9378(93)90339-k. PMID 8357043
- [Background] Saunders S, Bocking A, Challis J, Reid G. Effect of Lactobacillus challenge on Gardnerella vaginalis biofilms. Colloids Surf B Biointerfaces. 2007 Apr 1;55(2):138-42. doi: 10.1016/j.colsurfb.2006.11.040. Epub 2006 Dec 9. PMID 17234391
- [Result] Wilson JD, Shann SM, Brady SK, Mammen-Tobin AG, Evans AL, Lee RA. Recurrent bacterial vaginosis: the use of maintenance acidic vaginal gel following treatment. Int J STD AIDS. 2005 Nov;16(11):736-8. doi: 10.1258/095646205774763081. PMID 16303068
- [Result] Andersch B, Forssman L, Lincoln K, Torstensson P. Treatment of bacterial vaginosis with an acid cream: a comparison between the effect of lactate-gel and metronidazole. Gynecol Obstet Invest. 1986;21(1):19-25. doi: 10.1159/000298923. PMID 3485071
- [Result] Holley RL, Richter HE, Varner RE, Pair L, Schwebke JR. A randomized, double-blind clinical trial of vaginal acidification versus placebo for the treatment of symptomatic bacterial vaginosis. Sex Transm Dis. 2004 Apr;31(4):236-8. doi: 10.1097/01.olq.0000118423.20985.e7. PMID 15028938
- [Result] Boeke AJ, Dekker JH, van Eijk JT, Kostense PJ, Bezemer PD. Effect of lactic acid suppositories compared with oral metronidazole and placebo in bacterial vaginosis: a randomised clinical trial. Genitourin Med. 1993 Oct;69(5):388-92. doi: 10.1136/sti.69.5.388. PMID 8244360
- [Derived] Tidbury F, Brulhart G, Muller G, Pavicic E, Weidlinger S, Eichner G, von Wolff M, Stute P. Effectiveness and tolerability of lactic acid vaginal gel compared to oral metronidazole in the treatment of acute symptomatic bacterial vaginosis: a multicenter, randomized-controlled, head-to-head pilot study. BMC Womens Health. 2025 Jan 6;25(1):7. doi: 10.1186/s12905-024-03513-1. PMID 39762879